CLINICAL TRIAL: NCT03406624
Title: Epigenetic and Molecular Biomarkers in Chronic Low Back Pain and Modic Changes
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital, Akershus (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Kjersti Storheim, Head of FORMI, Oslo University Hospital
Other Study IDs: 2015/697
Record Dates: First submitted 2017-12-20; First posted 2018-01-23 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Low Back Pain
Keywords: Modic changes; biomarkers; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Spinal fusion with modic changes: Patients scheduled for surgery with lumbar spinal fusion with procedures involving moderate to extensive removal of the disc, and with modic changes seen on MRI at the actual level for surgery
  Interventions: Procedure: Biopsy
- Spinal fusion without modic changes: Patients scheduled for surgery with lumbar spinal fusion with procedures involving moderate to extensive removal of the disc, but with no modic changes seen on MRI at the actual level for surgery
  Interventions: Procedure: Biopsy
- Disc herniation surgery with modic changes: Patients scheduled for disc herniation surgery, and with modic changes seen on MRI at the actual level for surgery
  Interventions: Procedure: Biopsy
- Disc herniation surgery without modic changes: Patients scheduled for disc herniation surgery, but with no modic changes seen on MRI at the actual level for surgery
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsies will be taken from disc and / or endplates during elective lumbar fusion surgery or disc herniation surgery (endplate biopsy is omitted in disc herniation surgery)

SUMMARY:
In the present study the investigators aim to examine the presence of bacteria in the disc and Modic Changes (MCs) (bone). A prospective study with 1-year follow-up of two patient populations undergoing elective spinal surgery (spinal fusion or disc herniation surgery) will be conducted. Patients previously operated on at index level will also be included, and evaluated as sub-groups.

The following tissues are collected: dermis, sub-fascial tissue, nucleus pulposus, annulus fibrosus, and endplates. Endplate biopsies are only performed in patients undergoing fusion surgery.

All tissue samples undergoing culturing should be processed within 4 hours of sampling. The time for sampling and culture processing are noted for each sample. Details are available in a published Method article.

For each tissue sample, bacterial growth is recorded and identified at species level. Initially, the microbiologist grades the plates as "no growth", "possible contamination", and "significant growth".

Possible contamination means that the bacteria may be derived from the environment and can be introduced at any step from the sample is taken to the analyses in the laboratory.

The investigators will perform direct 16S rDNA Sanger sequencing on all frozen tissue samples.

Other broad metagenomic methods will also be considered, e.g., nanopore or Illumina sequencing.

Since C. acnes is considered the main pathogen in this setting, the investigators will also use a specific quantitative PCR on all samples.

The investigators will also use whole genome sequencing on C. acnes isolates for phylogenetic analyses to compare isolates found in samples from the same patient.

Based on cultivation alone, many samples will be clearly graded as "significant growth" or "no growth". Before unblinding, sensitivity analyses will be done after such "possible contamination" has been re-categorized as "significant growth" or "no growth" based on PCR and histological findings".

Microbiologists,the pathologist and clinicians are blinded until end of study.

Blood-samples are collected to characterize gene expression patterns and related markers.

DETAILED DESCRIPTION:
Planned analyses

Primary analyses:

MC1 vs. control (significant growth from disc, yes/no)

MC2 vs. control (significant growth from disc, yes/no)

Exploratory subgroup analyses:

MC1 and MC2 in previously operated vs. control (significant growth from disc, yes/no)

Large MCs vs. control (significant growth from disc, yes/no). Large MCs are defined as MCs with volume ≥ 25 % of vertebral body volume or height > 50 % of vertebral body height.

MC1 and MC2 vs. control in fusion group (significant growth from vertebral body biopsy, yes/no). Vertebral body biopsies are not performed in the disc herniation group.

Statistics and power:

The main aim of this study is to investigate if the proportions of patients with significant bacterial growth from perioperative disc biopsies differ between cases (MC1 patients or MC2 patients) vs controls without MCs. The null hypothesis is that there is no difference between cases and controls. The alternative hypothesis is that there is a difference.

The sample size calculation is based on previously published data and a pre-specified relevant difference in proportions of bacterial growth among cases vs. controls

The investigators calculated the sample size using a two-sided Pearson's chi-squared test. For the primary analysis, with two primary endpoints, the investigators aim to achieve 80 % power to detect a difference in bacterial growth in 25 % of cases with MC1 or MC2 vs. 5% of controls. Due to multiple testing the investigators use Bonferroni correction (alfa 0.025). The investigators therefore plan to analyze at least 60 cases with MC1, 60 cases with MC2 and 60 controls.

The MC2 sample is likely to become larger than n = 60, since the investigators recruit MC1 and MC2 patients consecutively and MC2 is more common than MC1.

The investigators will consider performing statistical sensitivity analysis where samples with possible contamination and positive PCR ("possible significant growth") are recategorized as positive bacterial growth.

The investigators will also consider sensitivity analyses with categorization of patients (positive/negative bacterial growth) depending on results from endplate, dermis and subfascia.

The primary endpoint will be analyzed with a logistic regression model with bacterial growth (positive/negative) as the outcome and group (MC1 or MC2 vs. control) as the main explanatory variable.

After fitting the model, the model-predicted marginal probabilities of positive bacterial findings will be estimated for both groups. The effect measure will be the difference between the two probabilities, and will be reported with a 95 % confidence interval and a P-value for the null hypothesis of a zero difference. The standard error of the difference will be estimated using the delta method.

The exploratory and sensitivity analyses will be carried out with the same model, after replacing outcome and main explanatory variable as appropriate. The subgroup analysis of previously operated will be carried out by adding previously operated as an interaction term between groups, and previously operated as covariates in the logistic model. A significant coefficient for the interaction term will indicate a subgroup effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery with lumbar spinal fusion with procedures involving moderate to extensive removal of the disc or disc herniation surgery (for cases: MC seen on MRI at the actual level for surgery, for controls: no MC seen on MRI at the actual level for surgery)
* LBP in the area below the 12th rib and above the gluteal folds
* Age > 18 years
* Written informed consent

Exclusion Criteria:

* Antibiotic treatment within the preceding one month before surgery
* Use of glucocorticoids the preceding month before surgery
* Small dots (i.e. <= 5 mm or height <10% of vertebra) are not included for any cases or control group
* Unwilling to participate
* Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from orthopaedic outpatient clinics at four university hospitals. They will be asked for participation after being scheduled for surgery with lumbar spinal fusion with procedures involving moderate to extensive removal of the disc (i.e. transforaminal lumbar interbody fusion (TLIF), posterior Lumbar Interbody Fusion (PLIF)) or or disc herniation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Microbiological analysis (aerob, anaerob cultivation) | During surgery
Histopathology and PCR | During surgery
Gene expression profiling | During surgery

SECONDARY OUTCOMES:
Oswestry disability index | Pre surgery, 3 and 12 months postoperatively
  The Oswestry Disability Index (ODI) provides the level of self-reported impairment of activity of daily living due to low back pain. There are 10 items in the ODI, each rated on a Likert scale from 0-5. The total range of possible scores is from 0 -50, which is converted to a percentage ranging from 0-100. The percentage of self-reported disability ranges from 0='no impairment' to 100='complete impairment'.
Roland and Morris Disability Questionnaire | Pre surgery, 3 and 12 months postoperatively
  The Roland Morris Questionnaire (RMQ) provides the level of self-reported impairment of activity of daily living due to low back pain. There are 24 items in the RMQ, each answered yes/no on a dichotomous questionnaire. All items answered with "yes" are summarized into a scale ranging from 0='no impairment' to 24='complete impairment'.
Low back pain | Pre surgery, 3 and 12 months postoperatively
  Self-reported level of low back pain, measured on a 0 to 10 Likert scale anchored by 0 indicating "no pain" and 10 indicating "unbearable pain".
Leg pain | Pre surgery, 3 and 12 months postoperatively
  Self-reported level of leg pain, measured on a 0 to 10 Likert scale anchored by 0 indicating "no pain" and 10 indicating "unbearable pain".
Health-related quality of life (EQ-5D) | Pre surgery, 3 and 12 months postoperatively
  EQ-5D, measuring patients health-related quality of life, have 5 dimensions: "Mobility", "Human Autonomy," "Current Daily Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 5 problem levels corresponding to patient response choices. A quality of life score is obtained according to the answers to the questionnaires.
Magnetic Resonance Imaging | Pre surgery and 12 months postoperatively (12 months postoperatively only for patients undergoing lumbar disc herniation surgery
  Magnetic Resonance Imaging (MRI): Sagittal T1- and T2 weighted images, axial T2 weighted images, sagittal short tau inversion recovery (STIR) images, sagittal fat-water separation images, sagittal diffusion weighted images (DWI), and sagittal T1 weighted DCE images (only if the patient can receive gadolinium injection). The same MRI protocol and the same type of 1.5 Tesla MRI scanners will be used at all study sites.
Blood samples | Pre surgery and 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Smeland, Professor, Study Director — Oslo University Hospital
Locations (4):
- Norway (4):
  - Haukeland University Hospital, Bergen
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital Ullevål, Oslo
  - Stavanger Universitetssjukehus, Stavanger

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rolfsen MP, Gammelsrud KW, Espeland A, Braten LC, Mjones SB, Austevoll I, Dolatowski FC, Arrestad MB, Toppe MK, Orlien IE, Holberg-Petersen M, Fagerland M, Zwart JA, Storheim K, Hellum C. Bacterial growth in patients with low back pain and Modic changes: protocol of a multicentre, case-control biopsy study. BMJ Open. 2024 May 6;14(5):e082244. doi: 10.1136/bmjopen-2023-082244. PMID 38719329